CLINICAL TRIAL: NCT01862848
Title: Topical Compounded Pain Creams And Pain Perception (TOPCAPP)
Acronym: TOPCAPP
Status: Completed | Type: Observational
Sponsor: Medimix Specialty Pharmacy, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Medimix Pharm-01
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Pain
Keywords: Topical Compounded Pain Creams and Pain Perception
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate the change in patient pain perception with the use of a topical compounded pain cream regimen.

DETAILED DESCRIPTION:
This is a prospective,observational,single center, open label study of patients that receive a combination topical compounded analgesic medication with no comparator group.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with an ICD9 code indicative of chronic pain.
* Participants must be starting a new regimen of topical therapy with multiple compounded agents.
* Participants must be expecting to receive therapy for at least 12 weeks.
* Participants must be between 18 and 65 years of age.
* Participants must be able to provide sound written and verbal informed consent.

Exclusion Criteria:

* Participants must not have prior hypersensitivity or adverse events to any of the components in the customized prescription.
* Participants must not be pregnant or breastfeeding women.
* Participants must not have a diagnosis of cancer within the past 5 years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with neuropathic or nociceptive chronic pain who are between 18 and 65 years of age prescribed a combination compounded topical analgesic.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Perceived pain changes | 12 Week Study [Baseline, 4,8, and 12 week evaluation]
  Minimal sample size of 60 persons(maximum n=150)with a diagnosis of chronic pain (n=30 neuropathic and n=30 nociceptive primary pain-type)to determine predictors of a 30% or greater reduction of pain scores evaluated by logistic regression analyses utilizing the Brief Pain Index scores.

SECONDARY OUTCOMES:
Quality of Life | 12 Weeks [Baseline,4,8, and 12 week evaluation]
  To evaluate the change in quality of life using the EuroQol-5D-3L survey.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Epstein, PharmD, Study Chair — Medimix Specialty Pharmacy
Locations (1):
- The Medimix Specialty Pharmacy, LLC, Jacksonville, Florida, United States

REFERENCES:
- [Background] Gureje O, Von Korff M, Simon GE, Gater R. Persistent pain and well-being: a World Health Organization Study in Primary Care. JAMA. 1998 Jul 8;280(2):147-51. doi: 10.1001/jama.280.2.147. PMID 9669787
- [Background] National Centers for Health Statistics, Chartbook on Trends in the Health Americans 2006, Special Feature: Pain. Available at: http://www.cdc.gov/nchs/data/hus/hus06.pdf. Accessed July 17,2012.
- [Background] Vorobeychik Y, Gordin V, Mao J, Chen L. Combination therapy for neuropathic pain: a review of current evidence. CNS Drugs. 2011 Dec 1;25(12):1023-34. doi: 10.2165/11596280-000000000-00000. PMID 22133325
- [Background] Chaparro LE, Wiffen PJ, Moore RA, Gilron I. Combination pharmacotherapy for the treatment of neuropathic pain in adults. Cochrane Database Syst Rev. 2012 Jul 11;2012(7):CD008943. doi: 10.1002/14651858.CD008943.pub2. PMID 22786518
- [Background] American Pain Foundation. Breakthrough cancer pain: mending the break in the continuum of care. J Pain Palliat Care Pharmacother. 2011;25(3):252-64. doi: 10.3109/15360288.2011.599920. PMID 21882979
- [Background] Flores MP, Castro AP, Nascimento Jdos S. Topical analgesics. Rev Bras Anestesiol. 2012 Mar-Apr;62(2):244-52. doi: 10.1016/S0034-7094(12)70122-8. PMID 22440379
- [Background] Barkin RL. Topical Nonsteroidal Anti-Inflammatory Drugs: The Importance of Drug, Delivery, and Therapeutic Outcome. Am J Ther. 2015 Sep-Oct;22(5):388-407. doi: 10.1097/MJT.0b013e3182459abd. PMID 22367354
- [Background] Clinical Pharmacology [database online]. Tampa, FL: Gold Standard, Inc., 2012. http://www.clinicalpharmacology.com